CLINICAL TRIAL: NCT05506670
Title: Disease Burden of RSV in Young Children in Primary Care
Brief Title: Disease Burden of RSV
Acronym: RSV ComNet III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL22_0703
Record Dates: First submitted 2022-08-12; First posted 2022-08-18 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-01

CONDITIONS: RSV Acute Respiratory Infection
Keywords: RSV infection; pediatrics; clinical burden; socio economic burden
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proved RSV infection (RSV positive patients (Experimental)
  Interventions: Other: Diagnostic test and phone call; Diagnostic Test: Diagnostic test
- suspected but not proved RSV infection (RSV negative patients) (Experimental)
  Interventions: Other: Diagnostic test and phone call; Diagnostic Test: Diagnostic test

INTERVENTIONS:
Other: Diagnostic test and phone call — Viral diagnostic test will be performed at inclusion. In case of RSV positive results, follow up phone calls will be scheduled at day 14 and day 30 to collect data.
Diagnostic Test: Diagnostic test — Viral diagnostic test will be performed at inclusion. In case of RSV negative result, no more intervention will be required.

SUMMARY:
Respiratory diseases are one of the leading causes of morbidity and mortality among young children, and respiratory syncytial virus (RSV) is the most common pathogen causing these respiratory diseases in this age group. RSV can present in the form of a variety of clinical syndromes, including upper respiratory tract infections, bronchiolitis, pneumonia, exacerbations of asthma and viral-induced wheeze. RSV is highly seasonal and occurs mostly during winter seasons in temperate climates. Sixty to seventy percent of all children experience an RSV infection before the age of one, and nearly all do so before the age of two.(

'Burden of disease' is a general term without a universally accepted definition and refers to the human and economic costs that result from poor health. RSV 'burden of disease' studies in young children (aged 0-4 years), have mostly been focused on the morbidity and mortality rates of RSV infections. The socio-economic burden of RSV infections in young children has been studied, however, a meta-analysis showed that of the 365,828 RSV disease episodes included in cost-analysis studies, only 27,286 (7.4%) focused on outpatient and emergency cases. To our knowledge, only two outpatient studies have prospectively investigated the clinical and socio-economic burden of laboratory confirmed RSV infections in young children; and both studies collected data in the early 2000s. More recently, one study has investigated the health care use, duration of illness and complications associated with RSV in a cohort of newborn infants. There is therefore a lack of knowledge on the clinical and socio-economic disease burden of RSV infections in young children in primary care.

Current treatment options for RSV infections are limited to supportive care. The only available antiviral monoclonal antibody (mAb) 'Palivizumab' is considered cost-effective for certain high-risk group infants and requires monthly injections during winter. New candidate RSV vaccines and mAbs (with longer half-life times) are in late-stage clinical trials. Therefore, accurate estimates of the burden of RSV infections, including in primary care, are crucial to better assess the overall impact RSV infections may have on the society.

ELIGIBILITY:
Inclusion Criteria:

1. Age <5 years
2. Consulting a primary care practitioner with symptoms of an acute respiratory infection (ARI)
3. Participation agreement of at least one of the two parents/legal guardians before intervention

Follow-up criterion

1) Sampled children with a lab-confirmed diagnosis of RSV.

Exclusion Criteria:

1. Signs of severity (moderate to severe respiratory distress, oxygen saturation SpO2 < 92%, dehydration, Glasgow < 13) for children < 3 month-old in emergency department
2. No consultation with a doctor in the previous 24 hours
3. Insufficient knowledge about the national language by the parents/legal guardians
4. Intellectual disabilities of the parents/legal guardians
5. Special personal circumstances in the family (based on the judgement of the primary care physician e.g. a recent death in the family)

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-02-24 (Actual); Study Completion 2024-02-24 (Actual)

PRIMARY OUTCOMES:
Clinical burden of RSV acute respiratory infections | Day 14
  Persistent symptomatology at D14
Clinical burden of RSV acute respiratory infections | Day 30
  Persistent symptomatology at D30

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre d'Investigation Clinique de Lyon- Groupement Hospitalier Est- Hospices Civils de Lyon, Bron, Rhone
  - Maison Médicale de l'Enfant, Écully, Rhone
  - Cabinet CAPELLI, Lyon, Rhone
  - Maison Médicale de l'Enfant, Écully, Rhône
  - Cabinet Bellemin, Villeurbanne, Rhône

IPD SHARING:
Plan to Share IPD: No